CLINICAL TRIAL: NCT02644564
Title: Early Clinical Examination and Ultrasonography Screening of Acute Soft Tissue Shoulder Injuries
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Martine Enger, MD, Oslo University Hospital
Other Study IDs: 2015/195
Record Dates: First submitted 2015-12-31; First posted 2016-01-01 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Soft Tissue Shoulder Injury; Rotator Cuff Tear
Keywords: Soft tissue shoulder injury; Rotator cuff tear; Ultrasonography
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasonography: Patients will undergo structured clinical examination and ultrasonography of both shoulders on the day of inclusion. They also fill out an injury registration form, Oxford Shoulder Score and QuickDASH. Follow-up at 3, 6 and 12 months will be identical, but without ultrasonography and injury registration form.
  Interventions: Other: Ultrasonography

INTERVENTIONS:
Other: Ultrasonography — One doctor does the clinical examination, another does ultrasonography. Both doctors and patient are blinded until results have been registered on written forms. The results are then disclosed to the patient and doctors in order to plan further treatment.

SUMMARY:
The purpose of the study is to determine whether the introduction of early ultrasonography screening will change the diagnostic spectrum of soft tissue shoulder injuries in patients aged forty years or more. We also want to study whether certain physical tests will be able to predict or rule out full-thickness tears of the rotator cuff (shoulder tendons) in the acute phase. Another purpose is to explore the course of soft tissue shoulder injuries over a year, as well as to compare the results to studies on the prevalence of rotator cuff full-thickness tears.

ELIGIBILITY:
Inclusion Criteria, all of the following:

* patient at Section for Orthopaedic Emergency, Oslo University Hospital
* living in the municipality of Oslo
* acute injury
* sudden onset of symptoms
* International Classification of Diseases (ICD) -10 S4-diagnosis (except injuries of middle and distal third of humerus and related soft tissue)
* no sign of acute injury on radiographs in two views, or successfully reduced dislocation without fracture
* turns up for follow-up appointment within 21 days of injury

Exclusion Criteria:

* patients that are incapable of giving and or receiving adequate information, or that cannot undergo a normal clinical investigation, due to for example language problems, level of consciousness, drugs, mental or emotional status or other
* patients that have undergone shoulder surgery during the last 6 months
* injury of both shoulders
* patients with neck-/shoulder problems or generalised muscle pain during the last three months before the injury
* other serious disease such as cancer, rheumatic disorders, haematological, neurological, endocrinological or gastrointestinal disease that according to the doctor's best clinical judgement makes participation or follow-up difficult
* does not want to participate

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients living in the municipality of Oslo that visit Section for Orthopaedic Emergency (Oslo skadelegevakt), Oslo University Hospital with an acute shoulder injury.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-10-05 (Actual); Primary Completion 2016-10-17 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Detection of full-thickness rotator cuff tear | Within 21 days of acute shoulder injury
  To explore the number of acute traumatic full-thickness tears in soft tissue injuries in the ≥ 40 population, and whether structured clinical examination is an adequate screening tool

SECONDARY OUTCOMES:
Oxford Shoulder Score (OSS) | Within one year of shoulder injury
  The OSS is a patient reported outcome score consisting of 12 items. It was developed for use in assessing the outcome of shoulder surgery, but is also used to assess non-surgical interventions. Each item is scored from 0 to 4, and the overall scores ranges from 0 to 48. The request for a licence to use the score was approved by Isis Outcomes on July 2nd 2015.
Shortened Disabilities of the Arm, Shoulder and Hand questionnaire (QuickDASH) | Within one year of shoulder injury
  QuickDASH is a patient reported outcome score consisting 11 of the original 30 items of the disabilities of the arm, shoulder and hand (DASH) questionnaire. Each item has five options, and the total score ranges from 0 - 100. The Norwegian translation used in the study is available at http://dash.iwh.on.ca/system/files/translations/QuickDASH_Norwegian.pdf

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ivar Brox, MD PhD, Study Chair — Oslo University Hosital
Locations (1):
- Section for Orthopaedic Emergency, Orthopaedic department, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Enger M, Schmidt M, Nordsletten L, Moosmayer S, Pripp AH, Melhuus K, Brox JI. Physical examination tests in the acute phase of shoulder injuries with negative radiographs: a diagnostic accuracy study. BMC Musculoskelet Disord. 2025 Jun 3;26(1):546. doi: 10.1186/s12891-025-08754-1. PMID 40462009